CLINICAL TRIAL: NCT00343876
Title: A Single Center, Double-Blind, Randomized Trial to Evaluate the Effects of Aspirin 325 mg + Clopidogrel 75 mg v. Aspirin 325 mg + Placebo on Plasma Concentration of C-Reactive Protein: The CATER Trial Protocol
Brief Title: Clopidogrel and Aspirin Together: The Effect on C-Reactive Protein Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi-Synthelabo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 128-012
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: hs-CRP; aspirin; clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel

INTERVENTIONS:
Drug: aspirin
Drug: clopidogrel

SUMMARY:
Inflammation is associated with worsening outcomes among individuals with CAD; C-reactive protein is a well-known marker of inflammation. Both healthy patients and those with a history of CAD who exhibit elevated CRP are at greater risk for cardiovascular events. Despite CRP's well- documented association with increased risk in the development and progression of CAD, the specific mechanism of elevated CRP in CAD is not known. One possible etiology includes a continuous prothrombotic process associated with CAD. Several studies demonstrate a link between platelet activation and inflammation. If thrombotic processes are involved in the mechanism of elevated CRP, antiplatelet therapy, including clopidogrel, could effectively reduce CRP. Preliminary studies have demonstrated a reduction of CRP with aspirin and a clear association between clopidogrel therapy and reduced CRP, however no randomized trials have been performed. We hypothesize that the proinflammatory effects of platelet activation may be inhibited with combined clopidogrel and aspirin therapy.

DETAILED DESCRIPTION:
The objective of this trial is to assess the effects of combined therapy of clopidogrel and aspirin versus placebo and aspirin on CRP in patients with known CAD.

Potential subjects already on stable aspirin and statin therapy will be randomized to clopidogrel vs. placebo in a I: 1 design. Participants will undergo study therapy for 3 months. Various laboratory parameters, including serum plasma concentration of CRP, will be assessed throughout the study. The primary endpoint is the effect of study therapy on CRP.

ELIGIBILITY:
Inclusion Criteria:

* Either gender > 18 years of age
* Documented coronary artery disease (CAD) of~ 70% documented lesion
* Must be taking 325 mg/day of aspirin (preferably Ecotrin)and a statin at least 4 weeks prior to enrollment
* The patient or legally authorized representative must sign a written informed consent, prior to the any procedure, using a form that is approved by the local Institutional Review Board
* Able to give informed consent

Exclusion Criteria:

* Documented sensitivity to aspirin or clopidogrel
* Uncontrolled hypertension as determined by the investigator
* Known bleeding disorder or increased risk of bleeding such as: severe hepatic, insufficiency, current peptic ulceration, proliferative diabetic retinopathy, history of bleeding diathesis or coagulopathy
* History of severe systemic bleeding such as: gastrointestinal bleeding, gross hematuria, intraocular bleeding, hemorrhagic stroke, intracranial hemorrhage
* Hospitalization for any MI or unstable angina in last 90 days
* Scheduled for a major surgery requiring prolonged study drug cessation (more than 4 weeks)
* Currently taking a thienopyridine agent (clopidogrel or ticlopidine), oral GP IIb/IIIa inhibitor, oral anticoagulant, or dipyridamole
* Pregnant and/or lactating women, and women of child bearing potential not using acceptable means of contraception. Women of childbearing potential must be using adequate measures of contraception (as determined by the investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period. Women of childbearing potential must have a negative pregnancy test at screen.
* Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the observation of the effect of aspirin + clopidogrel vs.
aspirin + placebo on CRP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Healthcare, LDS Hospital
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States